CLINICAL TRIAL: NCT05346978
Title: Effect of Consumption of a Lyophilized Nasturtium (Tropaeolum Majus L), on the Insulin Response, Lipid Profile, Antioxidant Capacity and Gene Expression in Pre-diabetic Subjects: Bogotá-Colombia
Brief Title: Nasturtium (Tropaeolum Majus L) Intake and Biochemical Parameters in Pre-diabetic Subjects in Bogota Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javeriana University (Other)
Collaborators: Leibniz Institute of Vegetable and Ornamental Crops (IGZ) (Unknown); University Medical Center Freiburg (Other)
Responsible Party: Principal Investigator, Valentina Guzman, Professor, Javeriana University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 7147
Record Dates: First submitted 2022-04-05; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Pre Diabetes
Keywords: Tropaeolum majus L.
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasturtium (NT) (Experimental): 5g freeze-dried nasturtium leaf powder ; Each participant was supplemented with 15 grams of freeze-dried nasturtium leaf powder (NT) or placebo (PLC) per wk during 4 wk. Each participant received 3 envelopes per wk with 5 g NT each or 3 g PLC. In total each participant was given 24 envelopes (12 NT and 12 PLC) packaged in the same way to be indistinguishable from each other. The participants were instructed to take three days at wk one NT or PLC envelope diluted in 300 ml (about 10.14 oz) in chilly water in a bottle provided for the study
  Interventions: Dietary Supplement: Nasturtium (Tropaeolum majus)
- Placebo (PLC) (Placebo Comparator): 3g collagen colored with green pigment used in the food industry; Each participant was supplemented with 15 grams of freeze-dried nasturtium leaf powder (NT) or placebo (PLC) per wk during 4 wk. Each participant received 3 envelopes per wk with 5 g NT each or 3 g PLC. In total each participant was given 24 envelopes (12 NT and 12 PLC) packaged in the same way to be indistinguishable from each other. The participants were instructed to take three days at wk one NT or PLC envelope diluted in 300 ml (about 10.14 oz) in chilly water in a bottle provided for the study
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nasturtium (Tropaeolum majus) — Freeze dried nasturtium (Edible flower)
  Arms: Nasturtium (NT)
Dietary Supplement: Placebo — collagen colored with green pigment used in the food industry
  Arms: Placebo (PLC)

SUMMARY:
Brassicaceae plant family have a high content of bioactive compounds such as e.g. glucosinolates (GSLs) and isothiocyanates (ICTs) associated, recently, with diabetes prevention. This research proposal has the intention of evaluating if the ingestion of freeze-dried nasturtium has a positive effect on the insulin response, lipid profile, oxidative stress biomarkers and gene expression of RESISTIN, GLUT 4, acetyl-CoA carboxylase-a (ACC), fatty acid synthase (FASN), NRF-2, NQO1, SFRXN1, glutathione peroxidase 2 (GPx-2), FOXO1, FOXO3 and FOXO6 in subjects with glucose intolerance.

DETAILED DESCRIPTION:
Epidemiological and animal studies have shown that consumption of fruits and vegetables decreases the risk of chronic diseases. Especially in T2D, the primary prevention is considered as a public health priority. Some studies show an inverse association between vegetables intake and T2D prevention, although the underlying mechanisms and the effect of individual antioxidant compounds are still unclear.

Brassicaceae plant family (e.g., broccoli, cabbage, brussels sprouts, watercress, Nasturtium, garden cress, kale, cauliflower), have a high content of bioactive compounds such as e.g. glucosinolates (GSLs), isothiocyanates (ICTs) and polyphenols, associated, recently, with diabetes prevention (18). Human studies in diabetic patients have shown that the consumption of broccoli sprouts powder (BSP) containing high concentration of the GLS sulphoraphane for 4 weeks decreases serum insulin concentration, homoeostasis model assessment of insulin resistance (HOMA-IR), LDL, inflammation and antioxidant markers. Besides sulphoraphane other GLSs have showed a protective effect in diabetes. Recently, mice fed with very high fat diet (VHFD) supplemented with 5% of moringa concentrate rich in benzyl isothiocyanate showed that moringa isothiocyanates (MICs) improved glucose tolerance and insulin signaling; reduced plasma leptin, resistin, cholesterol, IL-1β, TNFα, and lower hepatic glucose-6-phosphatase (G6Pase) gene expression. This evidence suggest that MICs could play a role in T2D prevention probably by inhibiting rate-limiting steps in liver gluconeogenesis resulting in direct or indirect increase in insulin signaling and sensitivity.

Recently in vitro studies in human and osteosarcoma hepatoma cells (HepG2 cells) stimulated with benzyl isothiocyanate (BITC) from Tropaeolum majus, show that this compound is able of 1) regulate the insulin signaling pathway, 2) down-regulate the gene and protein expression of gluconeogenic enzymes G6Pase and phosphoenol piruvatokinase (PEPCK) and 3) up-regulate the gene expression of antioxidant and phase II detoxification genes manganese superoxide dismutase (MnSOD), nuclear factor (erythroid derived)-like2 (NRF2), NAD(P)H dehydrogenase (quinone 1) (NQO1) and sulfiredoxin-1 (SFRXN1) (21). According with this evidence BITC could mimics the fasting state, in which insulin stimuli is absent and transcription factors remain in the nucleus modulating gene expression of their target genes, with the advantage of down-regulating gluconeogenesis instead of increase it suggesting that BITC could have a therapeutic role in the prevention or treatment of T2D.

Despite of strong evidence of 1) chronic inflammation as an underlying cause of T2D, and 2) high levels of oxidative stress under T2D conditions the use of ITC-rich foods as therapeutics in T2D remains virtually unknown. For that reason this research proposal has the intention of evaluating if the ingestion of freeze-dried nasturtium has a positive effect on the insulin response, lipid profile, oxidative stress biomarkers and gene expression of RESISTIN, GLUT 4, acetyl-CoA carboxylase-a (ACC), fatty acid synthase (FASN), NRF-2, NQO1, SFRXN1, glutathione peroxidase 2 (GPx-2), FOXO1, FOXO3 and FOXO6 in subjects with glucose intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 25-60 years, with a clinical diagnosis of glucose intolerance for at least six months.
* Body mass index (BMI) > 30 kg/m2. The BMI will be restricted to > 30 kg/m2 to reduce the variability in the lipid profile parameters, which frequently are normal in subject with normal BMI.
* Sign informed consent

Exclusion Criteria:

* Severe impairment of cardiac, hepatic or renal function.
* Gestation or lactation
* Use of insulin injection
* Pharmacotherapy with metformin or iDPP4, which alter insulin sensitivity or Glycaemia
* Consumption of antioxidant or vitamin supplements
* Consumption of estrogen or vitamin K-antagonists

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Glucose response | 4 weeks
  Fasting and postprandial blood glucose (mmol/L) was measured by the enzymatic colorimetric method (Beckman Coulter, CA, USA)
Lipid profile | 4 weeks
  total cholesterol (mmol/L), triglycerides level (mmol/L), High density lipoprotein cholesterol (mmol/L) and Low density lipoprotein cholesterol (mmol/L) were measured by enzymatic colorimetric analysis (Beckman Coulter, CA, USA).

SECONDARY OUTCOMES:
IR-HOMA | 4 weeks
  Homeostatic model assessment for Insulin Resistance was calculated with the formula (Basal Insulin (μU/L) x fasting blood glucose (mmol/L)/22.5)
Insulin | 4 weeks
  Insulin (uU/mL) was measured by chemiluminescent microparticle immunoassay (CMIA) (Abbott, IL, USA).
Castelli's risk index I and II | 4 weeks
  CT/HDL-c and LDL-c/HDL-c were calculated as cardiovascular risk factors parameters, at baseline and 4 weeks after treatment.
Oxidized LDL | 4 weeks
  OX-LDL (pg/mL). For quantify the concentration of serum oxidized LDL used ELISA kit (Novus Biologicals, USA)
Atherogenic Coefficient (AC) | 4 weeks
  non- HDLc)/ HDL-c were calculated as cardiovascular risk factors parameters, at baseline and 4 weeks after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Guzman, PhD, Principal Investigator — Pontificia Universidad Javeriana
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahadoran Z, Mirmiran P, Hosseinpanah F, Rajab A, Asghari G, Azizi F. Broccoli sprouts powder could improve serum triglyceride and oxidized LDL/LDL-cholesterol ratio in type 2 diabetic patients: a randomized double-blind placebo-controlled clinical trial. Diabetes Res Clin Pract. 2012 Jun;96(3):348-54. doi: 10.1016/j.diabres.2012.01.009. Epub 2012 Feb 9. PMID 22325157
- [Background] Bahadoran Z, Tohidi M, Nazeri P, Mehran M, Azizi F, Mirmiran P. Effect of broccoli sprouts on insulin resistance in type 2 diabetic patients: a randomized double-blind clinical trial. Int J Food Sci Nutr. 2012 Nov;63(7):767-71. doi: 10.3109/09637486.2012.665043. Epub 2012 Apr 26. PMID 22537070
- [Background] Carter P, Gray LJ, Troughton J, Khunti K, Davies MJ. Fruit and vegetable intake and incidence of type 2 diabetes mellitus: systematic review and meta-analysis. BMJ. 2010 Aug 18;341:c4229. doi: 10.1136/bmj.c4229. PMID 20724400
- [Background] Dinkova-Kostova AT, Kostov RV. Glucosinolates and isothiocyanates in health and disease. Trends Mol Med. 2012 Jun;18(6):337-47. doi: 10.1016/j.molmed.2012.04.003. Epub 2012 May 10. PMID 22578879
- [Background] Gomez-Martinez S, Diaz-Prieto LE, Vicente Castro I, Jurado C, Iturmendi N, Martin-Ridaura MC, Calle N, Duenas M, Picon MJ, Marcos A, Nova E. Moringa oleifera Leaf Supplementation as a Glycemic Control Strategy in Subjects with Prediabetes. Nutrients. 2021 Dec 24;14(1):57. doi: 10.3390/nu14010057. PMID 35010932
- [Background] American Diabetes Association Professional Practice Committee. 3. Prevention or Delay of Type 2 Diabetes and Associated Comorbidities: Standards of Medical Care in Diabetes-2022. Diabetes Care. 2022 Jan 1;45(Suppl 1):S39-S45. doi: 10.2337/dc22-S003. PMID 34964876
- [Background] Platz S, Kuhn C, Schiess S, Schreiner M, Kemper M, Pivovarova O, Pfeiffer AF, Rohn S. Bioavailability and metabolism of benzyl glucosinolate in humans consuming Indian cress (Tropaeolum majus L.). Mol Nutr Food Res. 2016 Mar;60(3):652-60. doi: 10.1002/mnfr.201500633. Epub 2015 Dec 28. PMID 26610401
- See also: Nasturtium (Tropaeolum majus L.) contains high concentrations of benzylglcosinolate. We found that a hydrolysis product of benzyl glucosinolate-the benzyl isothiocyanate (BITC)-modulates the intracellular localization of the transcription factor Forkhead — http://doi.org/10.1371/journal.pone.0162397